CLINICAL TRIAL: NCT06430346
Title: Exercise Prehabilitation for Locoregional Esophageal Cancer: A Pilot Study
Brief Title: Exercise Prehabilitation for Locoregional Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23121
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise prehabilitation (Experimental): In this trial participants will participate in an exercise program for 5 to 17 weeks, varying with treatment plans. Participants will receive resistance training equipment and participate in resistance training sessions twice per week (approximately 30-45 minutes per session). A Fitbit device will be provided to monitor step counts.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Physical activity and resistance training

SUMMARY:
The purpose of the study is to examine the feasibility and acceptability of exercise "prehabilitation" for patients preparing for esophageal cancer resection (removal).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven locoregional esophageal cancer (LEC)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Treatment plan including neoadjuvant chemoradiation therapy and surgical resection
* Ability to read and speak English

Exclusion Criteria:

* Regular engagement in resistance training (2x/week targeting all major muscle groups)
* Screen failure for exercise safety based on PAR-Q
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease
* Recent fracture or acute musculoskeletal injury that precludes ability to participate in resistance training safely
* Numeric pain rating scale of 7 or more out of 10
* Myopathic or rheumatologic disease that impacts physical function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Retention | Up to 11 weeks
  The number of participants who complete T0 and T1 measures.

SECONDARY OUTCOMES:
Exploratory outcomes and changes | Up to 17 weeks
  The number of participants who demonstrate improvements in exploratory outcome measures.
Clinical and treatment outcomes | Up to 17 weeks
  Chi-square testing will be used to determine if there's a difference in perioperative outcomes between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Parker, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States